CLINICAL TRIAL: NCT00824785
Title: REAL 3 : A Randomised Open-labelled Multicentre Trial of the Efficacy of Epirubicin, Oxaliplatin and Capecitabine (EOX) With or Without Panitumumab in Previously Untreated Advanced Oesophago-gastric Cancer
Brief Title: REAL3 Trial of Efficacy of EOX With/Without Panitumumab in Previously Untreated Adv OG Cancer
Acronym: REAL3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor David Cunningham, Head GI & Lymphoma Units, Royal Marsden NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR3024
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Oesophago-gastric Cancer
Keywords: epirubicin; oxaliplatin; capecitabine; panitumumab
MeSH Terms: interventions — Epirubicin; Oxaliplatin; Capecitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A EOX (Active Comparator): EOX chemotherapy (epirubicin, oxaliplatin and capecitabine)
  Interventions: Drug: epirubicin, oxaliplatin, capecitabine (EOX)
- Arm B EOX + panitumumab. (Active Comparator): EOX chemotherapy with the addition of panitumumab 9mg/kg every 21 days
  Interventions: Drug: EOX + panitumumab

INTERVENTIONS:
Drug: epirubicin, oxaliplatin, capecitabine (EOX) — epirubicin 50mg/m(2) IV on day 1 oxaliplatin 130mg/m(2) IV on day 1 with hydration capecitabine 1250mg/m(2)/day PO in two divided doses continuously from days 1-21
  Arms: Arm A EOX
Drug: EOX + panitumumab — epirubicin 50mg/m(2) IV on day 1 oxaliplatin 100mg/m(2) IV on day 1 with hydration capecitabine 1000mg/m(2)/day PO in two divided doses continuously from days 1-21 panitumumab -9 mg/kg every 21 days
  Arms: Arm B EOX + panitumumab.

SUMMARY:
To determine whether adding panitumumab, an antibody against the epidermal growth factor receptor (EGFR), to standard chemotherapy with epirubicin, oxaliplatin and capecitabine (EOX), improves the duration of survival of patients with advanced stomach and oesophageal cancer.

DETAILED DESCRIPTION:
Multicentre phase III, open labelled, randomised controlled trial. Randomisation will be 1:1 Arm A EOX and Arm B EOX + panitumumab. There will be a pilot phase II study of which the first 200 patients will be randomised and the primary endpoint for interim analysis will be when these patients have completed 6 months follow-up

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified inoperable locally advanced or metastatic adenocarcinoma or undifferentiated carcinoma of the oesophagus, oesophago-gastric junction, or stomach.
* Slides of tumour tissue should be available for centralised EGFR staining
* Uni-dimensionally measurable disease (CT or MRI as per RECIST).
* No prior chemotherapy including previous adjuvant chemotherapy
* No prior radiotherapy including adjuvant radiotherapy. Patients receiving palliative radiotherapy to sites of disease that are not measurable may be eligible and should be discussed with the Chief Investigator.
* Male/female patients aged ≥18 years.
* WHO Performance status 0, 1 or 2.
* Patients should have a projected life expectancy of at least 3 months.
* Completion of baseline quality of life questionnaire (EORTC QLQ C30).
* Adequate cardiac function; formal measurement of left ventricular ejection fraction is only required if clinically indicated.
* Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5x109/l; white blood cell count ≥ 3x109/l; platelets ≥ 100x109/l; haemoglobin (Hb) ≥ 9g/dl (can be post-transfusion).
* Adequate renal function: calculated creatinine clearance ≥50ml/minute.
* Adequate liver function: serum bilirubin ≤1.5x ULN; ALT/AST ≤2.5x ULN; ALP ≤3x ULN (in the absence of liver metastases). If liver metastases are present, serum transaminases ≤5x ULN are permitted.
* Written informed consent must be obtained from the patient before any study-specific procedures are performed (see Section 12.0).

Note: Epidermal growth factor receptor (EGFR) positivity by immunohistochemistry will not be required for study entry. Slides obtained from previously collected paraffin embedded archived specimens will be collected centrally for EGFR staining. A multivariate analysis will then be performed to exclude any effects of EGFR status on outcome measures

Exclusion Criteria:

* Tumours of squamous histology.
* Patients with locally advanced oesophageal cancer suitable for definitive chemoradiotherapy.
* Documented or symptomatic brain metastases and/or central nervous system metastases or leptomeningeal disease.
* Previous chemotherapy or radiotherapy. See Inclusion criteria for note regarding palliative radiotherapy.
* Any major surgery within 4 weeks prior to the start of study treatment.
* Any prior treatment with an EGFR signal transduction directed therapy.
* Treatment with non-permitted medication.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, uncontrolled cardiac dysrhythmia, or myocardial infarction within the last 12 months. Patients with any history of clinically significant cardiac failure are excluded from study entry.
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan.
* Known peripheral neuropathy >Grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible).
* Lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, or inability to take oral medication (administration of capecitabine by naso-gastric or jejunostomy feeding tube is permitted).
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Known hypersensitivity to panitumumab, components of the EOX regimen, or any of the constituents of these agents.
* Known positive tests for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or chronic active hepatitis B infection.
* Other clinically significant disease or co-morbidity which may adversely affect the safe delivery of treatment within this trial.
* Female patients who may be pregnant or breastfeeding. Potential female patients of childbearing potential must have a negative pregnancy test within 7 days prior to randomisation, or have had amenorrhea for more than 2 years.
* Patients of child-bearing potential not consenting to use adequate contraceptive precautions or abstinence during the course of the study and for 6 months after the last study drug administration for females, and 1 month for males.
* Any other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix).
* Treatment with another investigational agent within 30 days of commencing study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2008-05; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Early termination
  Study closed early due to lack of efficacy

SECONDARY OUTCOMES:
response rate, toxicity, quality of life and PFS | Early termination
  Study closed early due to lack of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Prof Cunningham, David, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Bournemouth, Bournemouth
  - St Luke's Guildford, Guildford
  - Royal Liverpool, Liverpool
  - Royal Marsden NHS Foundation Trust, London
  - Clatterbridge Oncology Centre, Metropolitan Borough of Wirral
  - Newcastle, Newcastle
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Smyth EC, Vlachogiannis G, Hedayat S, Harbery A, Hulkki-Wilson S, Salati M, Kouvelakis K, Fernandez-Mateos J, Cresswell GD, Fontana E, Seidlitz T, Peckitt C, Hahne JC, Lampis A, Begum R, Watkins D, Rao S, Starling N, Waddell T, Okines A, Crosby T, Mansoor W, Wadsley J, Middleton G, Fassan M, Wotherspoon A, Braconi C, Chau I, Vivanco I, Sottoriva A, Stange DE, Cunningham D, Valeri N. EGFR amplification and outcome in a randomised phase III trial of chemotherapy alone or chemotherapy plus panitumumab for advanced gastro-oesophageal cancers. Gut. 2021 Sep;70(9):1632-1641. doi: 10.1136/gutjnl-2020-322658. Epub 2020 Nov 16. PMID 33199443
- [Derived] Waddell T, Chau I, Cunningham D, Gonzalez D, Okines AF, Okines C, Wotherspoon A, Saffery C, Middleton G, Wadsley J, Ferry D, Mansoor W, Crosby T, Coxon F, Smith D, Waters J, Iveson T, Falk S, Slater S, Peckitt C, Barbachano Y. Epirubicin, oxaliplatin, and capecitabine with or without panitumumab for patients with previously untreated advanced oesophagogastric cancer (REAL3): a randomised, open-label phase 3 trial. Lancet Oncol. 2013 May;14(6):481-9. doi: 10.1016/S1470-2045(13)70096-2. Epub 2013 Apr 15. PMID 23594787